CLINICAL TRIAL: NCT00134433
Title: Endothelial Modulation With L-Arginine in Patients Undergoing Angiogenic Therapy (EMAT): A 2x2 Factorial Trial
Brief Title: Endothelial Modulation for Angiogenic Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Marc Ruel MD MPH FRCSC, Dr., Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: NA5163
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease, Diffuse; Coronary Artery Disease, Deemed Inoperable
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: intramyocardial VEGF angiogenesis (at a dose of 2 mg)
Drug: oral L-arginine supplementation (at a dose of 6 g/day)

SUMMARY:
Coronary artery disease is the single most important killer of Canadians. Despite major advances in therapy, there is still a significant proportion of patients identified with the disease who die of it because current treatment approaches cannot effectively palliate their condition. A new treatment modality called therapeutic angiogenesis has appeared on the clinical research scene during the last five years; this approach recreates the natural processes of new blood vessel formation that is observed during growth and development in every human being. It is an extremely potent and promising modality, but so far the results of clinical trials in patients have been equivocal.

One reason for the limited efficacy observed thus far with therapeutic angiogenesis may rest in that factors produced by the lining of the coronary arteries themselves are essential for angiogenic substances to take effect in the heart muscle of patients with severe coronary artery disease. These same patients, however, virtually all have, as a result of their disease, marked dysfunction of their coronaries and therefore fail to produce these factors in adequate quantities. This hypothesis has been verified with extensive animal data by the investigators of this research, where a swine model of coronary disease was shown to severely inhibit the action of angiogenic growth factors. If one wants angiogenesis to work, a means of improving the function of the coronary lining of patients with severe ischemic heart disease must be identified and its effects evaluated in order to allow for angiogenic substances to exert their action towards successful revascularization of the heart muscle.

An amino acid called L-arginine has repeatedly been shown to markedly improve function of the coronary artery lining in patients with ischemic heart disease when administered regularly over a period of several months. This research will therefore test, in the form of a randomized clinical trial, whether this concomitant approach can make angiogenesis effective in patients with advanced coronary disease, by allowing for the action of growth factors to take place in the heart. If this approach is successful, as is anticipated, angiogenesis will constitute an effective modality for the treatment of coronary artery disease, not only in patients with advanced, severe involvement unamenable to any other form of cardiac therapy such as coronary artery bypass grafting, but even perhaps in all patients with coronary artery disease in need of revascularization. The goal of this investigation towards the making of a new, revolutionary, safe and efficacious modality for the treatment of the number one killer disease of Canadians is in complete agreement with the primary objective of the Heart and Stroke Foundation of Canada.

DETAILED DESCRIPTION:
The EMAT trial tests the hypothesis that the concomitant treatment of chronic endothelial dysfunction in patients undergoing angiogenic therapy can make angiogenesis clinically effective. This is achieved with a 2x2 factorial, double-blind, placebo-controlled randomized trial of intramyocardial vascular endothelial growth factor (VEGF) angiogenesis at a dose of 2 mg and of adjunct endothelial modulation therapy using oral L-arginine supplementation at a dose of 6 g/day in patients undergoing surgical perivascular angiogenic therapy. The study involves surgical angiogenesis techniques similar to those previously used and reported to be clinically safe by the principal investigator and collaborators. Patients with a diffusely disease left anterior descending (LAD) coronary artery have this artery grafted with an internal thoracic artery in either its proximal or distal portion (according to what is felt by the surgeon to be most optimal as per usual practice). The segment of the LAD that is not directly bypassed (i.e. either the proximal portion if a distal bypass is performed by the surgeon or the distal portion if a proximal bypass is performed) is treated by the surgeon with VEGF angiogenesis or placebo injections. Other coronary arteries in need of bypass grafting are grafted as per usual practice, using arterial grafts. Patients are therefore randomized to one of four groups at the time of coronary artery bypass grafting:

* growth factor (VEGF) angiogenesis along the diffusely diseased, non-directly bypassed LAD segment + L-arginine oral supplementation;
* placebo "angiogenesis" along the diffusely diseased, non-directly bypassed LAD segment + L-arginine oral supplementation;
* growth factor (VEGF) angiogenesis along the diffusely diseased, non-directly bypassed LAD segment + placebo oral supplementation; and
* placebo "angiogenesis" along the diffusely diseased, non-directly bypassed LAD segment + placebo oral supplementation.

The angiogenesis treatment consists either of the injection of 2 mg (divided in 10 injections of 200 μg each) of plasmid DNA encoding for the VEGF165 gene or of 10 x 1 ml injections of a sterile physiologic saline solution in the myocardial territory and septum along the diffusely diseased, non-directly bypassed LAD segment. Other myocardial territories are concomitantly revascularized with arterial coronary bypass grafts.

The EMAT trial's primary end-points relate to objective myocardial perfusion indices and contractility of the intervened anterior myocardial portion, respectively measured with cardiac positron-emission tomography (PET) by using the investigational radioisotope 13-N ammonia, and by RNA or echocardiography. Using 13-N PET, collateral-dependent blood flow and ischemic zone size are measured in a double-blind fashion by a single observer at baseline and at 3 months. To better delineate the actual effects of angiogenic therapy, baseline perfusion scans are obtained 3 to 5 days after the operative procedure in order to account for the potentially confounding effect of CABG on myocardial perfusion to the proximal and distal anterior and septal territories. The functional, secondary end-points of the EMAT trial consist of clinical outcomes including major adverse cardiac events (MACE), freedom from angina, and angina class.

ELIGIBILITY:
Inclusion Criteria:

* Severe chronic angina
* Multi-vessel coronary artery disease
* Diffusely diseased left anterior descending coronary artery (LAD)
* At least 18 years of age at the time of written informed consent

Exclusion Criteria:

* Pregnancy, lactation, or any child-bearing potential
* Patients who are candidates for percutaneous transluminal coronary angioplasty (PTCA) or stenting
* Severe left ventricular dysfunction (ejection fraction < 30%)
* Threatened proximal coronary occlusion or unstable angina
* Recent myocardial infarction (< 1 month)
* Chronic renal failure (serum creatinine > 130 µmol/L)
* Hepatic insufficiency (Child-Pugh Class C)
* Clinically significant valvular heart disease
* Personal history of neoplasia
* Abnormal serum prostate-specific antigen (PSA), bowel neoplasia screening questionnaire, or updated mammography report (if female) - any test not performed within the last 6 months will be conducted prior to confirmation of eligibility
* Family history of cancer (i.e. ≥ 2 first-degree relatives)
* History of diabetic retinopathy
* Latent herpes infection
* Schizophrenia
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-11; Primary Completion 2007-03 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Blood flow to ischemic zone at 6 months compared to baseline: Persantine Ammonia Perfusion PET done at baseline prior to discharge from hospital and repeated at 3 months post intervention
Echocardiogram done at baseline prior to discharge from hospital and repeated at 3 months post intervention
Freedom from angina recurrence: Study participant interview and Seattle Angina Questionnaire administered (3 months, 6 months, 1 year). Results compared from preoperative baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ruel, MD MPH FRCSC, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- Division of Cardiac Surgery, University of Ottawa Heart Institute, Ottawa, Ontario, Canada